CLINICAL TRIAL: NCT05738512
Title: Medial Flap Coblation Turbinoplasty Versus Submucous Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFM-IRB: R.22.09.1853
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inferior Turbinate Hypertrophy
Keywords: Inferior turbinate; turbinoplasty; submucous resection; medial flap; coblation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial Flap Coblation Turbinoplasty (Active Comparator)
  Interventions: Procedure: Medial Flap Coblation Turbinoplasty
- Submucous Resection (Active Comparator)
  Interventions: Procedure: Submucous Resection

INTERVENTIONS:
Procedure: Medial Flap Coblation Turbinoplasty — Reduction of the inferior turbinate to manage inferior turbinate hypertrophy
  Arms: Medial Flap Coblation Turbinoplasty
Procedure: Submucous Resection — Submucous Resection
  Arms: Submucous Resection

SUMMARY:
Both submucous resection and medial flap coblation turbinoplasty are equally effective and safe in relieving nasal obstruction and enabling optimal volume reduction with preservation of function of the inferior turbinate. Coblation turbinoplasty has superior outcomes in terms of better healing and less bleeding, postoperative pain and crusting. Medial flap turbinoplasty is a simple, minimally invasive easy to learn procedure with low morbidity and excellent long-lasting results.

DETAILED DESCRIPTION:
This prospective, randomized, comparative surgical trial was conducted in the Department of Otorhinolaryngology, Mansoura University, Egypt, over a period of 2 years (March 2020 - March 2022). The study included 90 adult patients with chronic nasal obstruction due to inferior turbinate hypertrophy, and not responding to the usual medical treatment (intranasal corticosteroid therapy for at least 3 months).

Patients with other causes of nasal obstruction such as chronic rhinosinusitis, sinonasal tumours and nasal septal deflections were excluded from the study. Additionally, patients with history of previous nasal surgeries were also excluded. All patients of the study (n=90) received prior medical treatment in the form of decongestants and intranasal corticosteroids with no improvement.

Patients of the study were randomly allocated into two groups using block randomization method: coblation medial flap turbinoplasty group (n=45), and submucous resection (SMR) group (n=45). The patients were blind to the procedure they had. Informed written consents were obtained from all participants (n=90), and the study was approved by the Mansoura Faculty of Medicine Institutional research board (MFM-IRB: R.22.09.1853).

All patients (n=90) were subjected for detailed history taking with special focus on the nasal symptoms.

Additionally, an objective assessment for the nasal airways was performed before and after surgery by rigid nasal endoscopic examination without using nasal decongestants. The inferior turbinate grading system that was applied by Camacho et al was adopted in the current study. It was classified into 4 grades: grade 1 (inferior turbinate occupying 0%-25% of total airway space), grade 2 (occupying 26%-50% of total airway space), grade 3 (occupying51%-75% of total airway space), grade 4 (occupying 76%-100% of total airway space).

Operative techniques:

All surgeries were performed under general anaesthesia. Patients were prepped and draped in the standard fashion for endoscopic sinus surgery, and by using a zero-degree rigid nasal endoscope, under video imaging.

Submucous resection (SMR):

After infiltration of the inferior turbinate with 1 to 2 ml of 1% lidocaine with 1:100,000 epinephrine solution, an incision was done along the infero-medial surface of the turbinate extending from posterior to anterior. Medial and lateral mucosal flaps were then elevated, followed by resection of the turbinate bone. Then, flaps were returned back into position

Medial flap coblation turbinoplasty:

Turbinoplasty was performed using Coblation II surgery system (Smith and Nephew, USA) with EVAC 70 wand set to: ablation power 7 and coagulation power 3. After infiltration with 1 to 2 ml of 1% lidocaine with 1:100,000 epinephrine, inferior turbinate in-fracture was done by using a Cottle dissector. The mucous membrane as well as the soft tissues of the lateral side of the inferior turbinate were excised in an anterior to posterior direction using the coblation in ablation mode. The turbinate bone was then dissected from the medial mucosa (raising a medial flap), by a Cottle dissector. The bone was removed, and haemostasis was adequately achieved by using the coblation in the coagulation mode for bleeding points. The medial flap was then repositioned inferiorly and laterally to cover the remining expoNo nasal packing was performed in both groups (n=90). Patients were discharged home on the next postoperative day. Oral antibiotics (amoxicillin-clavulanic acid) were prescribed for one week. Saline nasal wash was prescribed for 2 - 3 weeks postoperatively. Follow up visits were planned on a weekly basis for one month, then after 3 months and 6 months.sed part of the inferior turbinate.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with chronic nasal obstruction due to inferior turbinate hypertrophy not responding to the conventional treatment; mainly intranasal steroid spray for 3 months duratoin.

Exclusion Criteria:

* Patients with other causes of nasal obstruction such as chronic rhinosinusitis, sinonasal tumours and nasal septal deflections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
improvement of nasal breathing | within 6 months after surgery
  subjectively assessed preoperatively and postoperatively by using the NOSE scale, objective assessment of the size of the inferior turbinate by endoscope. The inferior turbinate grading system that was applied by Camacho et al was adopted in the current study. It was classified into 4 grades: grade 1 (inferior turbinate occupying 0%-25% of total airway space), grade 2 (occupying 26%-50% of total airway space), grade 3 (occupying51%-75% of total airway space), grade 4 (occupying 76%-100% of total airway space).

SECONDARY OUTCOMES:
Intra-operative bleeding | during surgery
  it was assessed by using the Boezaart surgical field grading scale as the following: Grade 0: no bleeding 'cadaveric condition', Grade 1: minimal bleeding, no required suction, Grade 2:minimal bleeding, occasional suction is required, Grade 3: minimal bleeding, frequent suction is needed, surgical field is threatened by bleeding few seconds after removal of suction, Grade 4: bleeding is moderate, frequent suction is required and surgical field is threatened by bleeding immediately after removal of suction, Grade 5: bleeding is severe, persistent suction is needed and surgical field is severely threatened by bleeding which can't be controlled by suction
Post operative pain | within 10 days afte surgery
  it was assessed by visual analogue scale (VAS), where the patient was asked to score the pain from 1 to 10 and was graded as following; zero: no problem, 1-3: mild problem, 4-7: moderate problem, and 8-10: severe problem.
Intra-nasal crustations | within 3 months after surgery
  it was evaluated according to the endoscopic score of "Lund and Kennedy", as the following: Grade 0: Absence of crustations, Grade 1: Mild crustations: partially filling the nasal cavity, Grade 2: Severe crustations: fully filling the nasal cavity.
Post-operative healing | within 3 months after surgery
  it was was evaluated also as regard Lund and kennedy, as the following: Good: if there are minimal crustations, fast mucosal re-epithelization, patient feels recovered from nasal symptoms, no nasal synechiae, Moderate: mild to moderate degree of crustations, mucosal re-epithelization, patient feels relief of nasal symptoms, with nasal synechiae, Poor: severe crustations and nasal synechiae, delayed mucosal re-epithelization patient doesn't feel relief of nasal symptoms, persistent inflammations and infection

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University faculty of Medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Omura K, Nomura K, Takeda T, Yanagi N, Kuroyanagi H, Yanagihara T, Tanaka Y, Kojima H, Otori N. How I Do It: Inferior Turbinectomy: Modified Techniques for Submucosal Resection. Allergy Rhinol (Providence). 2021 Aug 9;12:21526567211034736. doi: 10.1177/21526567211034736. eCollection 2021 Jan-Dec. PMID 34408915
- [Result] Farmer SE, Eccles R. Chronic inferior turbinate enlargement and the implications for surgical intervention. Rhinology. 2006 Dec;44(4):234-8. PMID 17216738
- [Result] Cavaliere M, Mottola G, Iemma M. Comparison of the effectiveness and safety of radiofrequency turbinoplasty and traditional surgical technique in treatment of inferior turbinate hypertrophy. Otolaryngol Head Neck Surg. 2005 Dec;133(6):972-8. doi: 10.1016/j.otohns.2005.08.006. PMID 16360523
- [Result] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Result] Camacho M, Zaghi S, Certal V, Abdullatif J, Means C, Acevedo J, Liu S, Brietzke SE, Kushida CA, Capasso R. Inferior turbinate classification system, grades 1 to 4: development and validation study. Laryngoscope. 2015 Feb;125(2):296-302. doi: 10.1002/lary.24923. Epub 2014 Sep 12. PMID 25215619
- [Result] Boezaart AP, van der Merwe J, Coetzee A. Comparison of sodium nitroprusside- and esmolol-induced controlled hypotension for functional endoscopic sinus surgery. Can J Anaesth. 1995 May;42(5 Pt 1):373-6. doi: 10.1007/BF03015479. PMID 7614641
- [Result] Lund VJ, Kennedy DW. Quantification for staging sinusitis. The Staging and Therapy Group. Ann Otol Rhinol Laryngol Suppl. 1995 Oct;167:17-21. PMID 7574265
- [Result] Bergmark RW, Gray ST. Surgical Management of Turbinate Hypertrophy. Otolaryngol Clin North Am. 2018 Oct;51(5):919-928. doi: 10.1016/j.otc.2018.05.008. Epub 2018 Jul 18. PMID 30029923